CLINICAL TRIAL: NCT01612273
Title: The Effect of Triflusal on Peripheral Microcirculation Dysfunction: A Double-Blind, Randomized, Controlled, Crossover Study.
Brief Title: The Effect of Triflusal on Peripheral Microcirculation Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2011-0018
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Vasospastic Syndrome
Keywords: Vasospastic syndrome; Vascular dysregulation
MeSH Terms: interventions — triflusal; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disgren (Experimental): Dose: 300mg bid, Mode of administration: oral, Duration: from randomization to 6 week, crossover-design.
  Interventions: Drug: Triflusal
- Aspirin (Experimental): Dose: 150mg bid, Mode of administration: oral, from randomization to 6weeks, crossover-design.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Triflusal — Dose: 300mg bid, Mode of administration: oral, Duration: from randomization to 6 week, crossover-design.
  Other Names: Disgren®
  Arms: Disgren
Drug: Aspirin — Dose: 150mg bid, Mode of administration: oral, from randomization to 6weeks, crossover-design.
  Other Names: Astrix
  Arms: Aspirin

SUMMARY:
To explore the efficacy of triflusal in patients with symptomatic peripheral microcirculation dysfunction. Triflusal is a salicylate compound approved in several countries as antithrombotic agent and it additionally has vasodilatory effect. The hypothesis is to explore if there is a improvement of peripheral microcirculation by triflusal.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 70 years of age
* Diagnosed vasospastic syndrome with nailfold capillaroscopy (Fingertip is subjected to carbon dioxide at -15°C for 60 seconds. People found to have a blood-flow standstill of at least 12s in one or more capillaries were defined as having vasospasticity)
* More than seven points in 10-question interview provided by Nagashima et al.
* Written informed consent

Exclusion Criteria:

* Prior documented diabetes
* Overt peripheral artery disease
* Pregnant or nursing
* bleeding tendency
* Any contraindication of antiplatelet agent
* Thrombocytopenia (platelet < 100,000mm3)
* Chronic liver disease (ALT > 100 IU/L or AST > 100 IU/L) or renal dysfunction (creatinine > 4.0 mg/dl)
* Patients who can not stop to take aspirin

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - The amount of blood flow measured by finger doppler ultrasonography. The improvement of subjective symptom measured by questionaire. | 6 weeks
  Comparison of the PSV (peak systolic velocity) and EDV (end diastolic velocity) measured by finger doppler ultrasonography between disgren and aspirin groups after 6 weeks treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, severance hospital, Seoul, Seoul, South Korea